CLINICAL TRIAL: NCT01580150
Title: Effects of Berries on Postprandial Glycemic Responses to Sucrose and Starch
Brief Title: Effects of Berries on Post-meal Blood Sugar
Acronym: SOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 247032; 70035/09, 1087/31/2009 (Other Grant/Funding Number: Tekes)
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Blood Glucose, Postprandial; Blood Insulin, Postprandial; Hyperglycemia
Keywords: Berries; Starch; Sucrose; Glucose; Insulin; Postprandial
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Berry meal (Experimental): Carbohydrate meals with berries
  Interventions: Other: Berries
- Reference meal (Active Comparator): Carbohydrate meals without berries
  Interventions: Other: No berries

INTERVENTIONS:
Other: Berries — Meals containing starch (bread) or sucrose are consumed with berries (150 g) or berry nectars (300 mL).
  Arms: Berry meal
Other: No berries — Meals containing starch (bread) or sucrose are consumed without berries.
  Arms: Reference meal

SUMMARY:
The purpose of this study is to investigate whether berries are effective in lowering blood glucose and insulin responses to meals containing starch or sucrose.

DETAILED DESCRIPTION:
Berries are rich sources of various polyphenols which may be beneficial in the regulation of blood glucose. In vitro and animal studies have shown that polyphenols and polyphenol-rich extracts of foods, including berries, may inhibit digestion and absorption of carbohydrates and thereby suppress postprandial glycemia. However, current evidence on the effects of berries on postprandial glycemic responses in humans is limited.

The purpose of this study is to investigate the effects of berries on postprandial glycemic responses (blood glucose and insulin) to starch or sucrose in healthy subjects. It consists of five substudies each of which includes 2-4 meals with different berry species typically consumed in Finland and a reference meal without berries. The following combinations of carbohydrates and berries are studied:

* Studies 1-2: white wheat bread (starch) is consumed with several berry species
* Study 3: white wheat bread or rye bread is consumed with a mixture of berries
* Study 4: sugar (sucrose) is consumed with berries and berry nectars
* Study 5: a sugar-sweetened bakery product (starch + sucrose) is consumed with berries and berry nectar.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-28 kg/m2
* normal fasting plasma glucose

Exclusion Criteria:

* Smoking
* Diabetes or other chronic disease
* Antibiotic medication within the past 3 months
* Blood donation within the past month

Ages: 25 Years to 69 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | 0, 15, 30, 45, 60, 90, 120 minutes post-meal
Plasma insulin | 0, 15, 30, 45, 60, 90, 120 minutes post-meal

SECONDARY OUTCOMES:
Plasma free fatty acids | 0, 15, 30, 45, 60, 90, 120 minutes post-meal

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Törrönen, Dr, Principal Investigator — Senior Scientist
Locations (1):
- University of Eastern Finland, Kuopio, Finland

REFERENCES:
- [Derived] Torronen R, Kolehmainen M, Sarkkinen E, Poutanen K, Mykkanen H, Niskanen L. Berries reduce postprandial insulin responses to wheat and rye breads in healthy women. J Nutr. 2013 Apr;143(4):430-6. doi: 10.3945/jn.112.169771. Epub 2013 Jan 30. PMID 23365108
- [Derived] Torronen R, Kolehmainen M, Sarkkinen E, Mykkanen H, Niskanen L. Postprandial glucose, insulin, and free fatty acid responses to sucrose consumed with blackcurrants and lingonberries in healthy women. Am J Clin Nutr. 2012 Sep;96(3):527-33. doi: 10.3945/ajcn.112.042184. Epub 2012 Aug 1. PMID 22854401